CLINICAL TRIAL: NCT04686643
Title: A Multicenter, Randomized, Double-blind, Phase III Study to Evaluate the Efficacy and Safety of AGSAVI in Patients With Essential Hypertension Inadequately Controlled With AGLS
Brief Title: Phase III Study to Evaluate the Efficacy and Safety of AGSAVI in Patients With Essential Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGSAVI1705
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — levamlodipine; Valsartan; Indapamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): AGSAVI
  Interventions: Drug: AGSAVI
- Reference (Active Comparator): AGLS
  Interventions: Drug: AGLS

INTERVENTIONS:
Drug: AGSAVI — S-amlodipine, Valsartan, Indapamide
  Other Names: S-amlodipine, Valsartan, Indapamide
  Arms: Treatment
Drug: AGLS — S-amlodipine, Valsartan
  Other Names: S-amlodipine, Valsartan
  Arms: Reference

SUMMARY:
A phase 3 study to evaluate efficacy and safety of AGSAVI

DETAILED DESCRIPTION:
A randomized, double-blind, multicenter, phase 3 study to evaluate efficacy and safety of AGSAVI for Inadequately Controlled with AGLS

ELIGIBILITY:
Inclusion Criteria:

* Hypertension patient who satisfied below condition at Visit 1.

  * patient who takes antihypertensive drug

    * 140mmHg <= sitSBP <= 200mmHg
  * patient who doesn't take antihypertensive drug

    * 160mmHg <= sitSBP <= 200mmHg
* Hypertension patient who satisfied below condition at Visit 2.

  * 140mmHg <= sitSBP <= 200mmHg at Visit 2
  * 130mmHg <= sitSBP <= 200mmHg at Visit 2(In high-risk patients)

Exclusion Criteria:

* Patient who have received 4 or more antihypertensive drug
* Patient with 20mmHg of difference in sitSBP or 10mmHg of difference in sitDBP between 2 times of BP measuring at Visit 1
* Patient with sitDBP >= 120mmHg at Visit 1 or 2
* Patient with secondary hypertension

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in sitSBP at week 10 | 10 weeks

SECONDARY OUTCOMES:
Change from baseline in sitting diastolic blood pressure at week 4 and week 10 | week 4 and week 10
Change from baseline in sitting systolic blood pressure at week 4 | week 4
•Proportion of subjects achieving Blood Pressure control | week 4 and week 10

IPD SHARING:
Plan to Share IPD: No